CLINICAL TRIAL: NCT07094984
Title: Multicenter, Randomized, Open-label, Three-arm Study on the Efficacy of Fecal Microbiota Transplantation vs Probiotic Therapy vs Eubiotic-gut-microbiota-boosting Diet in Order to Antibiotic-resistant Bacteria (ARB) Decolonization From the Gastrointestinal Tract of Patients Colonized With Clinically Most Significant ARBs. Looking for a Strategy to Overcome the WHO Alarm on the Antibiotic Resistance "New Pandemic" Threat. STOP-ARB Study
Brief Title: Comparison of Three Interventions for Antibiotic-Resistant Bacteria (ARB) Decolonization From the Gastrointestinal Tract
Acronym: STOP-ARB3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Human Biome Institute S.A. (Industry); Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STOP-ARB3; 2022/ABM/03/00044/P/07 (Other Grant/Funding Number: Medical Research Agency)
Record Dates: First submitted 2025-07-29; First posted 2025-07-31 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-04

CONDITIONS: Drug Resistance, Bacterial; Antimicrobial Drug Resistance
Keywords: Fecal Microbiota Transplantation; FMT; Antibiotic-resistant bacteria decolonization; Eradication procedure; probiotic therapy; eubiotic diet
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: The study uses a parallel assignment design where participants are randomly allocated to one of three groups: fecal microbiota transplantation (FMT), probiotic therapy, or a eubiotic gut microbiota-stimulating diet. Each group receives its assigned intervention concurrently without crossover or switching, allowing direct comparison of the interventions' effects on antibiotic-resistant bacteria decolonization.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fecal Microbiota Transplantation (FMT) group (Experimental): Participants in the Fecal Microbiota Transplantation (FMT) arm receive antibiotic pre-treatment for five days (days 1-5), followed by bowel cleansing on day 6. FMT is then administered either orally in capsule form on day 7 (full dose) and continued with a prolonged capsule intake regimen from days 9 to 14, or via colonoscopy on days 7 and 14 if capsules cannot be taken. The FMT material is provided by the Human Biome Institute and aims to restore a healthy gut microbiota to facilitate decolonization of antibiotic-resistant bacteria. Patients in this arm are hospitalized during the treatment phase for close monitoring.
  Interventions: Other: Fecal microbiota transplantation (FMT)
- Probiotic therapy group (Experimental): Participants in the probiotic therapy arm receive bowel cleansing on day 6, followed by oral administration of a multistrain probiotic preparation from days 7 to 26. The probiotic contains 8 bacterial strains, including 4 Lactobacillus, 3 Bifidobacterium, and 1 Streptococcus strain, with a total daily dose of 450 billion live lyophilized bacteria (administered twice daily). The goal is to support gut microbiota modulation and promote decolonization of antibiotic-resistant bacteria. Treatment and monitoring are conducted on an outpatient basis.
  Interventions: Dietary Supplement: Probiotic Therapy
- Eubiotic gut microbiota boosting diet group (Experimental): Participants in the diet arm receive a scientifically formulated, eubiotic gut microbiota boosting diet aimed at promoting the natural restoration of healthy intestinal flora and supporting spontaneous decolonization of antibiotic-resistant bacteria. The dietary intervention begins after bowel cleansing on day 6 and continues daily for 38 days. Meals are prepared and delivered by a specialized catering service according to a standardized nutritional plan developed by clinical dietitians. The intervention is conducted in an outpatient setting, with patients receiving instructions, materials, and monitoring tools at treatment initiation
  Interventions: Other: Gut Microbiota Boosting Diet

INTERVENTIONS:
Other: Fecal microbiota transplantation (FMT) — FMT administered after antibiotic pre-treatment and bowel cleansing. Delivered either in capsule form or via colonoscopy to restore healthy gut microbiota and support decolonization of ARB.
  Other Names: FMT; Fecal Microbiota Capsules; Stool Transplantation; Human Biome Institute FMT
  Arms: Fecal Microbiota Transplantation (FMT) group
Dietary Supplement: Probiotic Therapy — Oral administration of a high-dose multistrain probiotic containing Lactobacillus, Bifidobacterium, and Streptococcus strains for 20 days following bowel cleansing.
  Other Names: Multistrain Probiotic Supplement; Gut Microbiota Support Supplement
  Arms: Probiotic therapy group
Other: Gut Microbiota Boosting Diet — A structured 38-day diet designed to promote eubiosis and support spontaneous ARB decolonization. Meals are tailored and delivered to patients based on clinical nutrition protocols.
  Other Names: Microbiota-Stimulating Diet; Dietary Modulation of Gut Flora; Eubiotic Diet
  Arms: Eubiotic gut microbiota boosting diet group

SUMMARY:
The aim of this research experiment is to evaluate the effectiveness of fecal microbiota transplantation (FMT) preceded by antibiotic pre-treatment versus probiotic therapy and a standard-of-care equivalent diet designed to stimulate the growth of eubiotic gut microbiota (an active comparator enhancing the ethical value of the study and increasing the chances of spontaneous decolonization of antibiotic-resistant bacteria (ARB) in the absence of any active intervention recommended by Scientific Societies) in the decolonization of bacteria with the most clinically significant antibiotic resistance mechanisms from the gastrointestinal tract of colonized patients.

This study addresses the urgent need highlighted by the World Health Organization (WHO) for new strategies to combat antibiotic resistance, aiming to prevent its progression into a global pandemic that could undermine the achievements of modern civilization.

Study Hypotheses:

* The decolonization rate of ARB bacteria in patients undergoing the intervention (FMT or probiotic therapy) is the same as in patients treated with standard-of-care (SoC) alone.
* The decolonization rate of ARB bacteria in the intervention groups (FMT or probiotic therapy) is at least 20 percentage points higher than in patients treated with the standard approach (diet).

The findings from this study may contribute to developing innovative microbiota-based therapies for the decolonization of antibiotic-resistant bacteria and help reduce the global burden of antibiotic resistance.

DETAILED DESCRIPTION:
The aim of this research experiment is to evaluate the effectiveness of three interventions for decolonization of antibiotic-resistant bacteria (ARB) from the gastrointestinal tract of colonized patients. The interventions include fecal microbiota transplantation (FMT), multistrain probiotic therapy preceded by antibiotic pre-treatment and bowel cleansing, and an eubiotic gut microbiota boosting diet as an active comparator. This approach addresses the urgent global need to develop new strategies against antimicrobial resistance, a growing threat predicted to cause millions of deaths annually by 2050 and significant economic impact.

This is an open-label, randomized, controlled experiment with a 2:1:1 allocation ratio (FMT:probiotic:diet). The total planned recruitment is approximately 360 adult patients documented to be colonized with clinically significant antibiotic-resistant bacterial strains, including carbapenem-resistant Enterobacteriaceae, multidrug-resistant Pseudomonas aeruginosa, Acinetobacter baumannii, vancomycin-resistant Enterococci (VRE), and methicillin-resistant Staphylococcus aureus (MRSA). Patients must meet defined inclusion and exclusion criteria ensuring safety and appropriateness for the interventions.

The FMT intervention involves administration of standardized fecal microbiota preparations in capsule form or via colonoscopy on specified days, preceded by a 5-day course of targeted antibiotics and bowel cleansing to reduce the existing gut microbial load. The probiotic arm receives a defined multi-strain probiotic preparation twice daily for 20 days following similar bowel cleansing. The diet arm follows a scientifically formulated diet designed to promote eubiosis, delivered daily for 38 days.

Study visits are conducted at screening, treatment initiation, and multiple follow-up points extending to six months post-intervention to monitor safety, efficacy, and long-term outcomes. Clinical assessments include medical history, physical examination, vital signs, and laboratory testing. Biological samples such as stool, urine, saliva, and blood are collected for microbiological and genomic analyses to evaluate colonization status and mechanisms of decolonization.

Sample size calculations, based on power analyses, aim to detect a clinically significant difference in decolonization rates among the groups, with 142 patients in the FMT arm and 71 patients in each comparator arm in the intention-to-treat population, accounting for anticipated dropout and screening failure rates.

This experiment is designed to provide robust data on the relative efficacy and safety of FMT, probiotic therapy, and dietary modulation in eradicating ARB colonization, potentially informing future clinical practices and public health policies to combat antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Documented intestinal colonization with antibiotic-resistant bacteria confirmed by at least two positive cultures (rectal swabs or, alternatively, stool cultures), with the last positive result obtained at least 28 days prior to the planned procedure;
* Documented colonization by one or more of the following bacterial strains:

  1. Carbapenem-resistant strains with confirmed resistance mechanisms, including MBL+ (NDM+, VIM+, or others), KPC+, OXA-48+, or phenotypic carbapenem resistance without identified genetic mechanism;
  2. Multidrug-resistant Enterobacteriaceae resistant to beta-lactams and other antibiotics, especially ESBL-producing strains, including Escherichia, Enterobacter, Klebsiella spp., and/or P. aeruginosa, A. baumannii (commonly associated with the ESKAPE group);
  3. Gram-positive bacteria such as Enterococcus faecalis, Enterococcus faecium, or other vancomycin-resistant enterococci (VRE), as well as Staphylococcus aureus strains resistant to methicillin (MRSA) and/or vancomycin;
* Absolute neutrophil count (ANC) in peripheral blood >500/μL within 3 days prior to FMT; In case of tandem or repeated FMTs and expected neutrophil decline, the ANC test should be repeated before each FMT if the interval exceeds 3 days.

For patients without expected neutropenia (<500/μL), the blood count remains valid for 28 days;

* Estimated life expectancy of at least 12 months;
* Ability to swallow large capsules (confirmed using a test capsule) or absence of contraindications to colonoscopy;
* No history of anaphylactic shock due to food allergies and ability to tolerate probiotic supplementation;
* Provision of written informed consent to participate in the study.

Exclusion Criteria:

* Lack of consent to participate in the study or inability to establish logical contact and obtain consent from an authorized representative;
* Absolute neutrophil count (ANC) < 500 cells/μL on the day of FMT (within 3 days prior) or predicted decline to this level within the next 2 days;
* Diagnosed HIV infection with CD4 lymphocyte count < 250 cells/μL;
* Active infection requiring antibiotic therapy on the day of FMT or planned antibiotic use during the first 7 days following FMT;
* Symptoms or radiological/endoscopic evidence of gastrointestinal mucosal damage within 7 days prior to FMT (e.g., ulceration, perforation, gastrointestinal bleeding) posing a risk of serious adverse events;
* Contraindications for FMT administration via upper or lower gastrointestinal tract routes (e.g., gastrointestinal perforation, anal atresia, lack of intestinal continuity, or other);
* Inability to undergo preparatory therapy (oral antibiotics: colistin, vancomycin, gentamicin and/or bowel cleansing agents) prior to FMT;
* Inability to swallow large capsules (confirmed with test capsules) or contraindications for colonoscopy;
* Severe food allergy with history of anaphylactic shock or inability to tolerate probiotics;
* Pregnancy or breastfeeding;
* Severe medical conditions contraindicating study protocol adherence as determined by the treating physician (e.g., severe heart failure precluding bowel cleansing due to risk of fluid overload or dehydration);
* Participation in another clinical trial and administration of an investigational drug or device within 3 months prior to randomization;
* Reluctance or inability to comply with protocol requirements, including any physical, mental, or social condition that may impair the participant's ability to adhere to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Complete decolonization of gastrointestinal antibiotic-resistant bacteria (ARB) | 60 days after completion of assigned intervention
  Proportion of participants achieving complete decolonization of ARB from the gastrointestinal tract, defined as at least two consecutive negative rectal swab cultures (or stool cultures), taken at least one day apart, at day 60 following completion of the eradication procedure. Bacterial resistance mechanisms include ESBL, CRE, VRE, and MRSA. If available, PCR confirmation of absence of resistance genes is required for final classification as eradicated.

SECONDARY OUTCOMES:
Complete decolonization of ARB at days 30, 90, and 180 | 30, 90, and 180 days post-intervention
  Proportion of participants with complete decolonization of gastrointestinal ARB, confirmed by at least two negative rectal swab or stool cultures taken at least one day apart, at days 30, 90, and 180 following the end of intervention. PCR confirmation of eradication is required when baseline colonization was confirmed by PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Klinika Hematologii, Transplantologii i Chorób Wewnętrznych, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Yes, individual participant data (IPD) will be shared with other researchers. Data sharing will be conducted only after the signing of a confidentiality agreement (non-disclosure agreement) to ensure the privacy and protection of participant information. Access to the data will be granted upon reasonable request and subject to approval by the study sponsor and ethics committee.